CLINICAL TRIAL: NCT06662409
Title: Support for Bereaved Friend and Family Caregivers of Cancer Patients
Brief Title: Support for Bereaved Cancer Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rebecca Lehto, Associate Professor, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R03CA282943 (NIH)
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Bereavement; Cancer; Caregiver; Grief
Keywords: nature-based intervention; meditation; bereavement support; grief; directed attention; quality of life; anxiety; depression; cancer caregiver
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nature-based healing meditation (NBHM) intervention (Experimental): 6 nature-based healing meditation (NBHM) auditory modules intervention
  Interventions: Other: Nature-based healing meditation (NBHM) intervention

INTERVENTIONS:
Other: Nature-based healing meditation (NBHM) intervention — 6 nature-based healing meditation (NBHM) auditory modules available via the study website to facilitate bereavement (grief) recovery and assessed on parameters of directed attention, grief, and QOL (including parameters of depression/anxiety)

SUMMARY:
Friend and family caregivers of recently deceased cancer patients experience acute bereavement following the death. Post death bereavement is an intense period of mourning that includes an unfolding of the grief process and is characterized by strong emotions and demands on cognitive resources to those who have put aside their own needs to support the dying patient with cancer. This research will test the feasibility and acceptability of a nature-based healing meditation (NBHM) intervention to support cancer caregivers' during the bereavement process.

DETAILED DESCRIPTION:
Bereaved friend and family caregivers have taken on the burden of end-of-life care for patients with cancer who die in hospice care at home. Bereavement can be emotionally devastating, especially to those who have put aside their own needs to support the dying individual. Supporting bereaved CGs' emotional health and general well-being is a critical need. The proposed pilot study will evaluate the acceptability and feasibility of a 6-week low-tech nature meditation intervention aimed at supporting bereaved caregivers' who are in the first 6 months since the patients' death. The intervention, based on the mutually supportive role that meditation practices and nature have been shown to promote wellbeing, will be developed capitalizing on the strengths of the research team's early intervention work involving patients with advanced cancer and their caregivers. For this single group longitudinal study, Aim 1 will focus on the development of 6 nature-based healing meditation (NBHM) auditory modules available via the study website to facilitate bereavement (grief) recovery and assessed on parameters of directed attention, grief, and QOL (including parameters of depression/anxiety).

The 2nd aim will then evaluate acceptability and feasibility of the 6-week program of both content and delivery methods (numbers eligible vs. number consented; numbers consented vs. numbers completed; number of weeks using the intervention) for the intervention modules. We will then conduct semi-structured interviews with a small diverse representative sample of caregivers to evaluate benefits, satisfaction, and challenges in more depth. Fifty-five home-based cancer caregivers who recently experienced the death of their patient will be recruited from Hospice of Michigan. Testing will occur at baseline (Time 1; study week 0), at the intervention end (Time 2; week 6), and (Time 3; study week 12). This research targets a supportive caregiver intervention that will be flexibly delivered on-line for use at the caregiver's convenience. Once feasibility and acceptability for this new intervention to support bereaved caregivers are addressed, a larger scale randomized control trial will be sought.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older; Able and willing to provide reflexology
* Able to speak and understand English
* Have access to a telephone
* Able to hear normal conversation
* Cognitively oriented to time, place, and person (determined via recruiter)

Exclusion Criteria:

* Unwilling to perform return demonstration with 90% accuracy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure | From baseline to the end of intervention at 12 weeks
  The 4-item Feasibility of Intervention Measure was developed for evaluating the success of feasibility, demonstrate encouraging psychometric properties. The items that are scored on a scale of 0 to 4 where 0 indicates "completely disagree," and 4 indicates "completely agree". Thus, the range for each scale extends from 0 - 16 with higher scores indicating higher feasibility and acceptability.
Acceptability of Intervention Measure | From baseline to the end of intervention at 12 weeks
  The 4-item Acceptability of Intervention Measure was developed for evaluating the success of acceptability, demonstrate encouraging psychometric properties. The items that are scored on a scale of 0 to 4 where 0 indicates "completely disagree," and 4 indicates "completely agree". Thus, the range for each scale extends from 0 - 16 with higher scores indicating higher feasibility and acceptability.
Attention Function Index | From baseline to the end of intervention at 12 weeks
  Directed attention will be assessed with the Attention Function Index, a 16-item self-rating scale that measures perceived effectiveness in daily tasks that require cognitive function. Items are scored on an 11-point Likert scale ranging from 0, indicating "not at all," to 10, indicating "extremely well or a great deal." Higher scores indicate better cognitive functioning.
Prolonged Grief 13-Revised | From baseline to the end of intervention at 12 weeks
  Grief (Bereavement) will be measured with the Prolonged Grief 13-Revised prolonged grief scale, Ongoing testing demonstrates that the measure is consistently reliable and a valid instrument for classifying less adaptive grief responses. Thirteen items to assess symptoms of prolonged grief disorder. Ten items are scored on a Likert-style scale from 1, "not at all," to 5 "overwhelmingly" to indicate how often that item describes how they are feeling. Three of the items assess whether the respondent had lost a significant other, how long ago the death occurred, and impairment associated with symptoms. Scores of 30 or greater on the symptom items indicate prolonged grief disorder (PGD), and were associated with poorer emotional and mental health as well as work and social adjustment difficulties.
PROMIS-29: Quality of life | From baseline to the end of intervention at 12 weeks
  The PROMIS profile instruments are a collection of profile short forms, where each form contains items from 1 of 7 primary PROMIS domains (emotional, social, and physical function, pain interference, fatigue, sleep disturbance, health satisfaction). PROMIS tools were developed to create psychometrically robust fixed-length short forms that can be used across trials and clinical conditions.
  The PROMIS-29 assesses each domain with 4 questions each. Items are on a 5-point Likert scale that ranges from 0 to 4.
Acceptability and Feasibility Tracking | From baseline to the end of intervention at 12 weeks
  participant numbers referred vs numbers eligible; numbers eligible vs. number consented; numbers consented vs. number completed; number of weeks using the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan State University College of Nursing, East Lansing, Michigan, United States